CLINICAL TRIAL: NCT05739578
Title: Experiences of patıent's prımary Caregivers With Tracheostomy Suctioning Before Discharge
Brief Title: Caregiver Experiences With Tracheostomy
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Yeliz Sapulu Alakan, lecturer, Uludag University
Other Study IDs: YSAlakan
Record Dates: First submitted 2023-02-02; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Tracheostomy; Care Giving Burden; Caregiver
Keywords: Tracheostomy; Suctioning; Caregiver
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to determine the experiences of primary caregivers of patients with tracheostomies on tracheostomy suctioning procedure. This is a semi-structured qualitative study.

DETAILED DESCRIPTION:
The study sample consisted of eleven (11) primary caregivers of patients with tracheostomies who were hospitalized in the otolaryngology clinic of a university hospital in a province located in the northwest of Turkey. This study was conducted using a semi-structured interview technique with the primary caregivers of the patients. Interviews were audio-recorded during the data collection procedure. The content of the audio recordings obtained during each interview was evaluated by the researchers using the content analysis method. The data were categorized, coded, and analyzed by creating themes and sub-themes. It was observed that the primary caregivers of the patients expressed fear, sadness, and anxiety during the suctioning procedure performed by healthcare professionals or themselves during their hospitalization. It was determined that caregivers need information on suctioning practice and insufficient knowledge on emergencies worries them as well.

ELIGIBILITY:
Inclusion Criteria:

* Being a caregiver of patients with tracheostomy over the age of 18
* Volunteer.
* Being the primary caregiver of the patient,
* Ability to communicate verbally
* Normal psychological state.

Exclusion Criteria:

* Being a caregiver of tracheostomy patients younger than 18 years of age
* Rejecting the voluntary event,
* Not being the primary caregiver of the patient,
* Inability to communicate verbally
* Having a psychological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eleven primary caregivers of patients who volunteered to participate in the study were included.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Experiences of patient's primary caregivers with tracheostomy suctioning before dıschange | Interviews with each caregiver whose patient's discharge was planned lasted an average of 33 minutes. Interviews with a total of 11 caregivers were completed in 3 months.
  A data collection form included 12 questions related to the sociodemographic characteristics of patients and their primary caregivers. The semi-structured interview questions were as follows;1) How did you feel when the nurse/physician performed suctioning from the tube in your patient's throat for the first time? What did you think? 2) How did you feel when you heard that this process should be continued at home? What do you think? What was your reaction? 3)How did you feel when you performed tracheal suctioning for the first time? 4) What was your reaction when you first heard that suctioning will be your responsibility at home? 5)Are there any different topics/details you want to share related to tracheostomy suctioning before discharge?

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz ŞAPULU ALAKAN, Principal Investigator — Uudag Universty
Locations (1):
- Bursa Uludag university, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, CSR
Time Frame: After the research is published
Access Criteria: It will be shared by researcher Yeliz ŞAPULU ALAKAN to be used in meta analysis or other research.

REFERENCES:
- [Result] Kun SS, Davidson-Ward SL, Hulse LM, Keens TG. How much do primary care givers know about tracheostomy and home ventilator emergency care? Pediatr Pulmonol. 2010 Mar;45(3):270-4. doi: 10.1002/ppul.21169. PMID 20146395
- [Result] Loerzel VW, Crosby WW, Reising E, Sole ML. Developing the Tracheostomy Care Anxiety Relief Through Education and Support (T-CARES) Program. Clin J Oncol Nurs. 2014 Oct;18(5):522-7. doi: 10.1188/14.CJON.522-527. PMID 25253106
- [Result] McCormick ME, Ward E, Roberson DW, Shah RK, Stachler RJ, Brenner MJ. Life after Tracheostomy: Patient and Family Perspectives on Teaching, Transitions, and Multidisciplinary Teams. Otolaryngol Head Neck Surg. 2015 Dec;153(6):914-20. doi: 10.1177/0194599815599525. Epub 2015 Aug 18. PMID 26286873
- [Result] Amar-Dolan LG, Horn MH, O'Connell B, Parsons SK, Roussin CJ, Weinstock PH, Graham RJ. "This Is How Hard It Is". Family Experience of Hospital-to-Home Transition with a Tracheostomy. Ann Am Thorac Soc. 2020 Jul;17(7):860-868. doi: 10.1513/AnnalsATS.201910-780OC. PMID 32267725
- [Result] Daraie S, Hasanvand S, Goudarzi F, Rassouli M. Gaining Experience Over Time: The Family Caregivers' Perception of Patients with a Tracheostomy in Home Care. Iran J Nurs Midwifery Res. 2021 Mar 5;26(2):137-143. doi: 10.4103/ijnmr.IJNMR_173_20. eCollection 2021 Mar-Apr. PMID 34036061